CLINICAL TRIAL: NCT03341819
Title: Comparative Study Between Retained and Non-retained Urinary Catheter in Total Knee Arthorplasty With Epidural Anesthesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Navamindradhiraj University (Other)
Responsible Party: Principal Investigator, Satit Thiengwittayaporn, Associate Professor, Navamindradhiraj University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: COA 126/2560
Record Dates: First submitted 2017-11-09; First posted 2017-11-14 (Actual); Last update posted 2019-11-25 (Actual); Status verified 2019-11

CONDITIONS: Postoperative Urinary Retention; Urinary Tract Infections; Epidural Anesthesia
MeSH Terms: conditions — Urinary Tract Infections | interventions — Arthroplasty, Replacement, Knee; Urinary Catheterization

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Retained Urinary Catheter (Active Comparator)
  Interventions: Procedure: Total knee arthroplasty; Procedure: Urinary Catheterization
- Non-retained Urinary Catheter (Experimental)
  Interventions: Procedure: Total knee arthroplasty

INTERVENTIONS:
Procedure: Total knee arthroplasty — A surgical procedure in which parts of the knee joint are replaced with artificial parts (prostheses)
Procedure: Urinary Catheterization — Urinary catheterization is a latex, polyurethane, or silicone tube known as a urinary catheter is inserted into a patient's bladder via the urethra. Catheterization allows the patient's urine to drain freely from the bladder for collection.
  Arms: Retained Urinary Catheter

SUMMARY:
The purpose of this study is to compare the prevalence of postoperative urinary retention between retained and non-retained urinary catheter in total knee arthorplasty with epidural anesthesia

ELIGIBILITY:
Inclusion Criteria:

* Primary osteoarthritis of knee who were scheduled for a primary total knee arthroplasty

Exclusion Criteria:

* History of renal disease
* History of urinary tract infection
* History of previous urinary tract surgery
* Benign prostatic hypertrophy
* Bilateral total knee arthroplasty
* Revision total knee arthroplasty
* Patients who need intraoperative monitoring of urine output

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 242 (Actual)
Dates: Start 2017-11-06 (Actual); Primary Completion 2019-04-05 (Actual); Study Completion 2019-10-25 (Actual)

PRIMARY OUTCOMES:
postoperative urinary retention | 6 hours after surgery and 6 hours after remove urinary catherter
  Patients who didn't void within 6 hours with suprapubic discomfort and had a urinary volume 400 mL or more confirmed by single intermittent catheterization

SECONDARY OUTCOMES:
urinary tract infection | 7 days after surgery
  An infection of the kidney, ureter, bladder, or urethra. The symptoms are burning with urination and having to urinate frequently and fever > 38° C. Urine culture shows a bacterial colony count of greater than or equal to ten to the fifth colony-forming units per mL of a typical urinary tract organism.

CONTACTS AND LOCATIONS:
Overall Officials: Satit Thiengwittayaporn, M.D., Principal Investigator — Department of Orthopaedics, Faculty of Medicine Vajira Hospital, Navamindradhiraj University
Locations (1):
- Navamindradhiraj University, Dusit, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Thiengwittayaporn S, Uthaitas P, Hongku N, Tunyasuwanakul R, Limphunudom P, Leelachiewchankul F. Indwelling urinary catheterization was unnecessary in non-drainage total knee arthroplasty: a randomized controlled trial. Arch Orthop Trauma Surg. 2021 Mar;141(3):469-476. doi: 10.1007/s00402-020-03677-z. Epub 2020 Nov 12. PMID 33180187